CLINICAL TRIAL: NCT02187315
Title: Induction Chemotherapy Followed By Chrono-chemotherapy Concurrent With Intensity-modulated Radiotherapy In The Treatment Of Locally Advanced Nasopharyngeal Carcinoma PhaseⅡClinical Randomized Study
Brief Title: Induction Chemotherapy Followed By Chrono-chemotherapy Concurrent With IMRT Of Locally Advanced NPC Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Feng Jing (Other)
Responsible Party: Sponsor-Investigator, Feng Jing, Guiyang Medical College, Guiyang Medical University
Organization: Guiyang Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20140501
Record Dates: First submitted 2014-05-15; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Induction Chemotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melodie group (Experimental): Induction chemotherapy followed by cisplatin chrono-chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Device: Chrono-chemotherapy pump:Melodie; Drug: induction chemotherapy; Drug: cisplatin chrono-chemotherapy; Radiation: intensity-modulated radiation therapy
- Routine-chemotherapy group (Other): Induction chemotherapy followed by cisplatin routine-chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Device: Routine intravenous drip; Drug: induction chemotherapy; Radiation: intensity-modulated radiation therapy; Drug: cisplatin routine-chemotherapy

INTERVENTIONS:
Device: Chrono-chemotherapy pump:Melodie
  Arms: Melodie group
Device: Routine intravenous drip
  Arms: Routine-chemotherapy group
Drug: induction chemotherapy
Drug: cisplatin chrono-chemotherapy
  Arms: Melodie group
Radiation: intensity-modulated radiation therapy
Drug: cisplatin routine-chemotherapy
  Arms: Routine-chemotherapy group

SUMMARY:
Comparing induction chemotherapy followed by cisplatin chrono-chemotherapy concurrent combined with intensity-modulated radiation therapy (chrono-chemotherapy group) with induction chemotherapy followed by cisplatin routine-chemotherapy concurrent combined with intensity-modulated radiation therapy (routine-chemotherapy group) in the treatment of locally advanced nasopharyngeal carcinoma, observing the adverse reaction and effects of two groups,expected chrono-chemotherapy group can achieve lower toxicity, improve the curative effect, for the treatment of nasopharyngeal carcinoma provides a more reasonable way.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of early cure Ⅲ - Ⅳ stage of patients with advanced nasopharyngeal carcinoma (according to the 2010 UICC staging criteria, T3-4, N0-3), no evidence of distant metastasis (M0). A measurable tumor lesions;
2. Karnofsky score≥70;
3. Age 18-70 years old, male or female;
4. No major organ dysfunction; Normal bone marrow hematopoietic function (white blood cell ≥4．0×109／L，platelet≥100×109 /L. hemoglobin ≥100g/L)，normal liver function (total bilirubin、alanine aminotransferase、 aspartate aminotransferase ≤1.5 times the upper limit of normal)，normal renal function (creatinine ≤1.5 times the upper limit of normal) electrocardiogram does not affect the normal treatment;
5. To understand this study and sign informed consent form.

Exclusion Criteria:

1. A distant metastasis;
2. Patients with physical or mental illness, and researchers think that patients can't fully or adequately understand the possible complications of this study;
3. Pregnancy (confirmed by serum or urine β-HCG test) or between lactation period;
4. Serious complications, such as uncontrollable hypertension, heart function failure, diabetes, etc.; 5.Who had received radiation and chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 5 year

SECONDARY OUTCOMES:
Number of Participants with curative effect | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Guiyang Medical College/The Affiliated Cancer Hospital of Guiyang Medical College/Guizhou Cancer Hospital, Guiyang, Guizhou, China